CLINICAL TRIAL: NCT00253045
Title: Motivating HIV+ Women: Risk Reduction and ART Adherence
Acronym: KHARMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Marcia McDonnell Holstad, DSN, FNP-BC, Principal Investigator, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00045905; 1R01NR008094-01A1 (NIH)
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: HIV; AIDS
Keywords: Motivational Interviewing; antiretroviral therapy; medication adherence; risk reduction behaviors; women; HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Motivational group (Experimental): Group counseling using motivational interviewing
  Interventions: Behavioral: Motivational groups

INTERVENTIONS:
Behavioral: Motivational groups — Motivational interviewing in group format

SUMMARY:
The purpose of this study is to determine if a group motivational interviewing based intervention will increase adherence to antiretroviral medications and use of risk reduction behaviors.

DETAILED DESCRIPTION:
Women are the fastest growing group of persons with AIDS. They are often diagnosed later in the disease, when antiretroviral therapy (ART) is strongly indicated. Currently ART involves the use of multiple medications that must be taken under strict conditions at regular time intervals up to as many as 4 different times a day. Some medications must be taken on an empty stomach, some with high fat food, some with low fat food, and all of these must be coordinated throughout the day. It is extremely important for patients to take ART exactly as prescribed and not miss any doses in order to reduce the amount of HIV virus in the bloodstream, increase the CD4 cell counts, prevent the serious consequences of AIDS, hospitalizations, and development of drug resistant strains. These regimen-related problems and the high care-taking burden placed on HIV+ women for their children and partners make near perfect adherence difficult to achieve. And, as women on ART begin to feel better and resume their normal activities, including sexual activities, adherence to behaviors that contribute to reducing the risk of spreading HIV (RRB), such as condom use and safe needle use in injection drug users becomes crucial. Researches have shown that only about 11% to 63% of HIV+ women use condoms consistently.

The primary purpose of this randomized controlled behavioral trial is to test the effect of a nurse led group motivational intervention for HIV+ women on adherence to ART and RRB. The secondary purpose is to examine the mediator effect of 3 variables that have been shown to be important in behavior change: self-efficacy, outcome expectancy, and personal goals. The Motivational Group + Usual Care (MG+UC) intervention builds on the usual care provided at the agencies and has Motivational Interviewing (MI) as a central component. It consists of 8 90 minute sessions, 1 week apart, led by a specially trained nurse, to motivate women to adhere to both ART and RRB. The intervention will be compared to an 8 session health promotion program (HPP+UC) that is led by a nurse health educator. These sessions will focus on nutrition, exercise, stress management, and women's health issues. These sessions will also be 90 minutes in length and meet weekly for 8 weeks. Both groups will receive beauty and pampering incentives such as beauty makeovers, skin care instruction, and massages after several of the sessions, as well as child care, transportation tokens, and monetary incentives of $10 for attendance at each of the first 4 groups and $15 for attendance at each of the last 4 groups. Snacks appropriate for ART and immune status will be supplied to the MG+UC group, and fruits, vegetables, and other nutritious snacks will be provided to the HPP+UC group. Groups will be held at AID Atlanta, the Infectious Disease Program of the Grady Health System, and at the Infectious Disease Clinic of Emory Crawford Long.

In order to be eligible to participate, the women must be HIV+, over 18 years of age, be on a new or different ART or have self-reported nonadherence to her current ART regimen, speak and understand English, and be mentally stable as determined by a screening assessment. All participants will complete a baseline assessment, and follow-up assessments immediately, 3, 6, and 9 months after the end of the group. Participants will be paid $25 for each assessment. We expect 300 women to be randomized and participate; pregnant women will not be excluded.

We hypothesize that the women who are randomized to the MG+UC group, will, on the immediate, 3, 6, and 9 month follow-up assessments have higher mean adherence rates to ART, report more frequent use of RRB, have higher CD4 counts, and lower mean viral loads than those randomized to the HPP+UC group. We also hypothesize that the effects of the intervention on adherence to ART and RRB will be brought about by higher mean levels of self-efficacy, more positive expected outcomes, and more specific and effective personal goals.

As noted above, MI forms the basis for the intervention. MI is a client-focused method of counseling used to help clients deal with ambivalence about changing behavior. MI principles include expressing empathy, developing discrepancy, rolling resistance, and supporting self-efficacy. It has been used primarily with individuals, but some MI groups have been described with substance users. Our application in a group format with HIV+ women is new and innovative.

All participants will receive the usual care plus either the Health Promotion Program or the Motivational Interviewing Intervention. How the usual care is administered varies by agency but in general for ART consists of prescription of new or different ART regimen based on established clinical criteria and guidelines by the Panel on Clinical Practices for Treatment of HIV infection, education about the medications (including actions, side effects, special requirements), setting up the medication schedule, and follow-up regarding medication taking. The usual RRB education includes information about risk reduction practices such as condom use, sexual practices, needle cleansing, and needle sharing. Depending on the agency, the usual care may be formalized and administered by health care providers, nurses, social workers, and/or health educators.

This innovative project is designed to promote adherence to both ART and RRB, something that has not been described so far in the literature. Adherence to ART promotes health and reduces infectiousness, including transmission of HIV from mother to fetus. Adherence to RRB reduces the spread of HIV. Thus, if effective, the intervention will promote health of HIV+ women and reduce the spread of HIV.

ELIGIBILITY:
Inclusion Criteria:

* Infected with HIV
* Be on a new or different antiretroviral medication regimen or self report non-adherence to antiretroviral medications
* Must be 18 years of age or older
* Female by birth
* Understand and speak English
* Be willing to complete a screening interview to further determine if you are able to take part in the study
* Be willing to follow study requirements and use a MEMS cap on one of your antiretroviral meds

Exclusion Criteria:

* Under 18 years of age
* Transgender
* Males
* HIV negative
* Do not understand or speak English
* Do not achieve a satisfactory score on the screening interview
* Diagnosed as actively psychotic, severely depressed, or pose a risk of harm to themselves or others since these women may not be emotionally capable of sitting through lengthy, potentially emotional group or assessment sessions, or may be disruptive to other participants

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2004-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Adherence to antiretroviral therapy | Baseline, 2 weeks, 3, 6, 9 months post intervention
  Self report questionnaires, Electronic drug monitoring caps (MEMS)
Use of Risk Reduction Behaviors | Baseline, 2 weeks, 3, 6, 9 months post intervention
  Questionnaires about risky sexual behaviors, and substance use behaviors
Clinical indicators | Baseline, 2 weeks, 3, 6, 9 months post intervention
  CD4 and HIV viral load lab results from medical records

SECONDARY OUTCOMES:
Self-Efficacy | Baseline, Immediate post follow-up, 3, 6, 9 months post intervention
Outcome Expectancy | Baseline, 2 weeks, 3, 6, 9 months post intervention
Personal Goals | Immediate post follow-up, 3, 6, and 9 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marcia McDonnell-Holstad, DSN,RN-C,FNP, Principal Investigator — Nell Hodgson Woodruff School of Nursing, Emory University; Bridget F. Jones, RN,MSN,BSEd, Study Director — Nell Hodgson Woodruff School of Nursing, Emory University
Locations (1):
- Nell Hodgson Woodruff School of Nursing, Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Holstad MM, DiIorio C, Magowe MK. Motivating HIV positive women to adhere to antiretroviral therapy and risk reduction behavior: the KHARMA Project. Online J Issues Nurs. 2006 Jan 31;11(1):5. PMID 16629499
- [Result] Holstad MM, DiIorio C, Kelley ME, Resnicow K, Sharma S. Group motivational interviewing to promote adherence to antiretroviral medications and risk reduction behaviors in HIV infected women. AIDS Behav. 2011 Jul;15(5):885-96. doi: 10.1007/s10461-010-9865-y. PMID 21165692
- [Result] Holstad MM, Diiorio C, McCarty F. Adherence, sexual risk, and viral load in HIV-infected women prescribed antiretroviral therapy. AIDS Patient Care STDS. 2011 Jul;25(7):431-8. doi: 10.1089/apc.2010.0331. Epub 2011 Jun 11. PMID 21663541